CLINICAL TRIAL: NCT02808910
Title: Nudging: How Small Changes in the Cafeteria of the Feiring Heart Clinic Can Result in a Healthier Food Choice.
Brief Title: A Small Nudge for Better Health Through Reduced Salt Intake, Increased Vegetable Intake, and Smaller Portion Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Collaborators: NIBIO - Norwegian Institute of Bioeconomy Research (Other); Norwegian University of Life Sciences (Other); Animalia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016/231300
Record Dates: First submitted 2016-05-03; First posted 2016-06-22 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Disease; Obesity
Keywords: behavior; food intake; salt; vegetables; portion size; weight loss; habits
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Behavior; Weight Loss; Habits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Salt nudge (Experimental): The following changes will be made in the cafeteria: Salt will be placed in a corner of the buffet, rather than on each dining table. Other spices, without sodium, will be provided on the table. A sign will be placed on the table that nudges participants to try the other spices. Food in the buffet that is high in salt will be labeled with a negative-appearing symbol, and food in the buffet that is low in salt will be labeled with a positive symbol.
  Interventions: Behavioral: Nudged to eat less added salt and more other seasonings; Behavioral: Nudged to avoid foods high in salt content, and to choose foods low in salt content
- Vegetable nudge (Experimental): The following changes will be made in the cafeteria: Names of the vegetable dishes in the buffet will be made more attractive. Signs will be placed with reminders to eat more vegetables. Signs will be placed with a visual indication of the percentage of a meal that should consist of vegetables.
  Interventions: Behavioral: Nudged to eat more vegetables
- Portion size nudge (Experimental): The following changes will be made in the cafeteria: Smaller plates will replace the regular plates. Verbal and visual nudges to reduce portion size will be given. Utensils for self-serving calorie-dense foods in the buffet will be smaller than normal.
  Interventions: Behavioral: Nudged to eat smaller portions; Behavioral: Nudged to eat less calorie-dense food
- Combined nudge (Experimental): All three nudges are combined in this intervention.
  Interventions: Behavioral: Nudged to eat less added salt and more other seasonings; Behavioral: Nudged to avoid foods high in salt content, and to choose foods low in salt content; Behavioral: Nudged to eat more vegetables; Behavioral: Nudged to eat smaller portions; Behavioral: Nudged to eat less calorie-dense food
- Control groups (No Intervention): No changes are made to the cafeteria, compared to the pre-study situation. One control group participates after each of the nudges to control for effects of time of the year.

INTERVENTIONS:
Behavioral: Nudged to eat less added salt and more other seasonings
  Arms: Combined nudge; Salt nudge
Behavioral: Nudged to avoid foods high in salt content, and to choose foods low in salt content
  Arms: Combined nudge; Salt nudge
Behavioral: Nudged to eat more vegetables
  Arms: Combined nudge; Vegetable nudge
Behavioral: Nudged to eat smaller portions
  Arms: Combined nudge; Portion size nudge
Behavioral: Nudged to eat less calorie-dense food
  Arms: Combined nudge; Portion size nudge

SUMMARY:
This study will investigate whether small changes (nudges) made in a cafeteria, where participants eat for 4 weeks, can improve their food behavior and health during the 4 weeks, and 6 weeks and 6 months after their stay. Half the participants will be exposed to one of four types of nudges (focused on reducing salt intake, increasing vegetable intake, reducing portion size, and a combination of these nudges), and half of the participants will eat in the cafeteria as it is currently, without modifications.

DETAILED DESCRIPTION:
A healthy diet is an important pillar for public health and for the prevention of several lifestyle diseases (e.g. obesity, cardiovascular diseases). However, diet choices are often not conscious choices. While it may help to make individuals more aware of healthy options for example through education or nutrition labels, it remains difficult for many to eat healthy. The food environment in which choices are made has an impact on the choice. Smart design of the food environment may help individuals to make a healthier choice, by nudging them towards the healthier alternative, while not limiting the availability of the less healthy choice.

This study tests how these 'nudges' can affect food behavior and health of participants in a 4-week rehabilitation course at Feiring Heart clinic. Nudges will be implemented in the cafeteria at the clinic.

Three types of nudges will be tested:

* Salt nudge: aims to reduce salt (sodium) intake. Salt will be less easily available in the cafeteria, and other spices (without sodium) will be made easily available. Food in the buffet that is either very high or very low in salt will be labeled.
* Vegetable nudge: aims to increase vegetable intake. Names of the vegetable dishes in the buffet will be made more attractive, signs will be placed with reminders to eat more vegetables, and with visual indications of the percentage of vegetables that should be part of a meal.
* Portion size nudge: aims to decrease portion size. Smaller plates will be provided, and utensils for self-serving calorie-dense foods in the buffet will be smaller than normal.
* One period will also combine all the nudges described above.

Outcomes include measures of food intake during the 4-week rehabilitation course, and whether food habits 6 weeks and 6 months after the 4-week course have changed, compared to before the course. BMI will be monitored during the 4-week period and self-assessed in the 6 months after. Physical activity habits will be considered during the entire experimental period, and satisfaction with the cafeteria food and service will be monitored throughout to assess whether the nudges impact customer satisfaction.

Results are expected to be transferable to other heart clinics, and cafeterias in other institutions.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be part of the 4 week rehabilitation course at the Feiring heart clinic
* Participants should be willing and able to complete the necessary registration of food choices, and the relevant questionnaires

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05-20 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change in BMI from start of intervention to end of intervention | Measured at baseline at day 0 of intervention and at completion of intervention at day 28 of intervention)
  BMI is measured, and change in BMI between day 0 and day 28 is used.
Change in dietary habits 1 | 6 weeks after the 4 week intervention period
  Habits are compared with habits as listed before the start of the 4 week intervention period. Done through an online survey.
Change in dietary habits 2 | 6 months after the 4 week intervention period
  Habits are compared with habits as listed before the start of the 4 week intervention period. Done through an online survey.

SECONDARY OUTCOMES:
Dietary choices in cafeteria 1.1 | Tuesday lunch meal during the first week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added
Dietary choices in cafeteria 1.2 | Thursday lunch meal during the first week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added
Dietary choices in cafeteria 2.1 | Tuesday lunch meal during the second week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added
Dietary choices in cafeteria 2.2 | Thursday lunch meal during the second week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added
Dietary choices in cafeteria 3.1 | Tuesday lunch meal during the third week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added
Dietary choices in cafeteria 3.2 | Thursday lunch meal during the third week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added
Dietary choices in cafeteria 4.1 | Tuesday lunch meal during the fourth week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added
Dietary choices in cafeteria 4.2 | Thursday lunch meal during the fourth week of the intervention
  Participants make photos of their meal including drinks, and register any condiments or seasoning added

OTHER OUTCOMES:
Customer satisfaction of the cafeteria through a survey | Once per week during the intervention, on day 3, 11, 18 and 25 of the intervention
  A short questionnaire is answered by those eating in the cafeteria, regarding their satisfaction with the food and the cafeteria, to check that the nudges do not impact customer satisfaction negatively. Focus is on quality of the food, the available choices, and satisfaction with the cafeteria layout/atmosphere and staff. The survey is completed once per week.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Dufseth, Principal Investigator — LHL Helse
Locations (1):
- LHL-klinikkene Feiring, Feiring, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wansink, B. & Sobal, J. Mindless eating: The 200 daily food decisions we overlook. Environment and Behavior. 2007, 39(1):106-123. 2007
- [Background] Rolls BJ. Plenary Lecture 1: Dietary strategies for the prevention and treatment of obesity. Proc Nutr Soc. 2010 Feb;69(1):70-9. doi: 10.1017/S0029665109991674. Epub 2009 Dec 3. PMID 19954563
- [Background] Rozin, P., Scott, S., Dingley, M., Urbanek, J.K., Jiang, H., Kaltenbach, M. Nudge to nobesity I: Minor changes in accessibility decrease food intake. Judgment and Decision Making, 2011, 6:323-332.
- [Background] Just, D.R. & Wansink, B. Smarter Lunchrooms: Using Behavioral Economics to Improve Meal Selection. Chocies Magazine. 2009, 24(3).
- [Background] van Kleef E, Otten K, van Trijp HC. Healthy snacks at the checkout counter: a lab and field study on the impact of shelf arrangement and assortment structure on consumer choices. BMC Public Health. 2012 Dec 12;12:1072. doi: 10.1186/1471-2458-12-1072. PMID 23231863